CLINICAL TRIAL: NCT06882278
Title: Efficacy and Safety of Pulsed Radiofrequency Combined With Platelet-Rich Plasma Applied to the Sphenopalatine Ganglion in Treating Episodic Cluster Headache: A Study Protocol for a Multi-Center, Prospective, Open-Label, Propensity Score Match Cohort Study
Brief Title: Pulsed Radiofrequency Combined With Platelet-Rich Plasma Applied to the Sphenopalatine Ganglion in Treating Episodic Cluster Headache
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: People's Hospital of Zhengzhou University (Other); Huadong Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Director of Department of Pain Management, Beijing Tiantan Hospital
Other Study IDs: KY 2023-263-03-05
Record Dates: First submitted 2025-03-12; First posted 2025-03-18 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Cluster Headache; Pain Management; Episodic Cluster Headache
Keywords: Episodic Cluster Headache; Pain management; Pulsed Radiofrequency; Platlet-rich Plasma
MeSH Terms: conditions — Cluster Headache; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pulse Radiofrequency combined with Platelet Rich Plasma: The pulse treatment generator will be set to the automatic pulsed radiofrequency mode, with a temperature of 42°C, pulse frequency of 2Hz, pulse width of 20ms and treatment duration of 360s. After removing the radiofrequency electrode, 2 ml of LP-PRP mixture will be injected slowly into the sphenopalatine ganglion. Additional analgesics will be administered for participants' comfort during and after the procedure. If the patients were not satisfied with the outcome after one month, other treatment options will be available.
- Pulse Radiofrequency alone: The pulse treatment generator will be set to the automatic pulsed radiofrequency mode, with a temperature of 42°C, pulse frequency of 2Hz, pulse width of 20ms and treatment duration of 360s. Patient from this group will not receive PRP injection.

SUMMARY:
Cluster headache (CH) is one of the most severe pain accompanied by ipsilateral autonomic symptoms such as lacrimation and conjunctival injection. CH can be categorized into episodic cluster headache (ECH), chronic cluster headache (CCH), and probable CH. Intervention for CH requires a multifaceted and early approach and varies due to the heterogeneity of patients, which makes it difficult to formulate appropriate treatment plan, and the minimally invasive interventional therapy between drug and surgical treatment is still worth looking forward to.

The pterygopalatine ganglion, also known as SPG, is a essential proportion in activation of cortical structures and plays an important role in the pathogenesis of CH attacks, which makes it the potential therapeutic target in drug-resistant CH. Percutaneous pulsed radiofrequency (PRF) at SPG is a minimally destructive treatment which shows efficacy, safety, and repeatedly efficacy for refractory CH. PRF is a reliable alternative with few neurological side effects and complications for patients who have not responded to conservative treatment. However, the long term pain relieve is not satisfying. Platelet-rich plasma (PRP) is an autologous blood-derived product of 3 times concentrated platelet above average levels, which contains many growth factors, cytokines, chemokine, and cell-adhesion molecules, therefore function in the activation and synthesis of healing process, tissue proliferation and regeneration. Researches by Michno etc. and Giaccari etc. have proved that PRP combined with PRF therapy may provide more effective outcome than PRF alone in treatment of neuralgia, but whether the combined therapy can improve the efficacy of CH treatment is not clear. ECH occurs in 90% of the CH patients. The investigators assume that PRP combined with PRF acting on SPG might have better therapeutic effect on ECH than PRF alone, by giving combined treatment or PRF therapy alone according to patients willingness, the investigators plan on conducting this prospective trail to compare the clinical efficacy and safety of PRP combined with PRF versus PRF alone.

ELIGIBILITY:
Inclusion Criteria:

1. The diagnosis of ECH is confirmed according to the diagnostic criteria of the International Classification of Headache Disorders third edition 3 (Table 2), and the patient is within five days of the current cluster period；
2. The patient's age is between 18 and 70 years;
3. Patients have had ≥2 bouts previously, ≥4 typical (treated or untreated) attacks per week and usual bouts should last 4 weeks;
4. The patient's pain condition remains the same after preventive therapy with drugs available in our hospital such as verapamil, topiramate, lithium or steroids, or there is a reduction of less than 50% in the intensity and frequency of headache attacks, the duration of each attack and the dosage of auxiliary analgesic drugs used.

Exclusion Criteria:

1. Have atypical features: absence of cranial autonomic symptoms, post-traumatic onset, cluster-tic syndrome;
2. Abnormalities in blood measurements, liver and kidney function, blood glucose, coagulation, electrocardiography or chest radiography;
3. Infection at the puncture site;
4. Previous mental illness;
5. Previous history of narcotic drug abuse;
6. Prior anticoagulant or antiplatelet therapy;
7. An implantable pulse generator;
8. Previous history of invasive treatments such as pterygopalatine ganglion radiofrequency thermocoagulation and chemical destruction;
9. Current pregnancy or breast feeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Suitable participants will be screened at the pain management centre of Department of Pain Management, Beijing Tiantan Hospital, Capital Medical University in Beijing, China; Department of Pain Management, Henan Provincial People's Hospital, Henan, China; Department of Pain Management, Huadong Hospital, Fudan University, Shanghai. to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 242 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2028-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
change in the weekly frequency of cluster headache attacks | At 1 week, 2 weeks, 3 weeks after the operation
  The overall mean change from baseline in the weekly frequency of cluster headache attacks across weeks 1 through 3

SECONDARY OUTCOMES:
change in the weekly frequency of cluster headache attacks | At 1day, 3days, 1week, 2weeks, 1month, 3months, 6months and 1year after the operation
  the overall mean change from baseline in the weekly frequency of cluster headache attacks
the percentage of patients with a reduction of at least 50% in the weekly frequency of cluster headache attacks | At 1day, 3days, 1week, 2weeks, 1month, 3months, 6months and 1year after the operation.
  the percentage of patients with a reduction from baseline of at least 50% in the weekly frequency of cluster headache attacks
the degree of pain | At 1day, 3days, 1week, 2weeks, 1month, 3months, 6months and 1year after the operation.
  the degree of pain during headache attacks (NRS scores)
the duration of each headache attack | At 1day, 3days, 1week, 2weeks, 3 weeks, 1month, 3months, 6months and 1year after the procedure.
  the duration of each headache attack
dose of auxiliary analgesic drugs | At 1day, 3days, 1week, 2weeks, 3 weeks, 1month, 3months, 6months and 1year after the procedure.
  the dose of auxiliary analgesic drugs taken
self-rated patient satisfaction | At 1day, 3days, 1week, 2weeks, 3 weeks, 1month, 3months, 6months and 1year after the procedure.
  the self-rated patient satisfaction, from 0 point for unsatisfied to 10 points for very satisfied.
WHOQOL-BREF | At 1day, 3days, 1week, 2weeks, 3 weeks, 1month, 3months, 6months and 1year after the procedure.
  the degree of patient satisfaction measured by WHOQOL-BREF (World Health Organization Quality of Life Questionnaire).
adverse events | At 1day, 3days, 1week, 2weeks, 3 weeks, 1month, 3months, 6months and 1year after the procedure.
  For intraoperative AEs, the occurrence of puncture pain, headache, dizziness, nausea, vomiting, facial haematoma and other effects will be recorded. For postoperative AEs, headache, dizziness, facial numbness and other effects will also be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes